CLINICAL TRIAL: NCT04295889
Title: Towards HOMe-based Albuminuria Screening: an Implementation Study Testing Two Approaches
Acronym: THOMAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Kidney Foundation (Other); E-Zorg B.V. / KPN Health (Unknown); Healthy.io Ltd. (Industry); Hessels+Grob (Unknown); Copernicus Interchange Technology B.V. (Unknown); Amphia Hospital (Other)
Responsible Party: Principal Investigator, dr. R.T. Gansevoort, Professor of Medicine, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LSHM17076-SGF
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Albuminuria
Keywords: albuminuria; chronic kidney disease; cardiovascular disease; population screening; home based; e-Health; app; hypertension; diabetes mellitus; hypercholesterolemia
MeSH Terms: conditions — Albuminuria; Renal Insufficiency, Chronic; Cardiovascular Diseases; Alzheimer Disease; Hypertension; Diabetes Mellitus; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A will receive an invitation for home based albuminuria screening using a more conventional urine collection device (known as "Peespot Test").
  Interventions: Diagnostic Test: Approach A (PeeSpot urine collection device).
- Group B (Active Comparator): Group B will receive an invitation for home based albuminuria screening using an app (internet application) and an ACR dipstick test (known as "ACR| EU Test").
  Interventions: Diagnostic Test: Approach B (ACR | EU Test kit).

INTERVENTIONS:
Diagnostic Test: Approach A (PeeSpot urine collection device). — The participant will receive the PeeSpot urine collection device (Hessels+Grob B.V., Deventer, The Netherlands), which consists of a holder containing a urine collection pad (consisting of hygroscopic material containing). The holder can be placed back into the tube and can be easily sent to the laboratory by mail. In this urine, albumin, creatinine, and the ACR will be measured in the laboratory of the Amphia hospital.
  Arms: Group A
Diagnostic Test: Approach B (ACR | EU Test kit). — The participant will receive the ACR | EU test kit (Healthy.io Ltd, Tel-Aviv- Yafo, Israel), which consists of a urine test strip, a urine cup, a color calibrator and instruction to download a smartphone application. The participants have to download the smartphone application according to the instructions included in the kit. Results will be directly shown to the participant in the app.
  Arms: Group B

SUMMARY:
Chronic Kidney Disease (CKD) is a worldwide major public health problem that is associated with an increased incidence of kidney failure and cardiovascular events, that lead a high burden for affected patients and high costs for society. Symptoms of CKD occur late, when kidney function drops to below 30%. At that time preventive measures will have only limited efficacy. Protein excretion in urine has increasingly been recognized as early marker of CKD, and is often associated with high blood pressure, diabetes, and/or high cholesterol levels. These are all important risk factors for progression of kidney and cardiovascular disease. Population screening for urinary protein loss could detect a considerable number of subjects with yet unknown risk factors for progressive kidney and cardiovascular disease who can benefit of early intervention. However, there is no validated method for population screening yet. The aim is to to develop a home based population screening for elevated urinary protein loss. Two screening methods will be investigated, and yield and cost-effectiveness of these screening methods will be evaluated

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a worldwide major public health problem that is associated with an increased incidence of kidney failure and cardiovascular disease (CVD). To tackle this burden, screening for CKD among the general population could be beneficial to allow early detection and treatment. In the last decades, elevated albuminuria has increasingly been recognized as an early marker of generalized vascular endothelial damage, that predicts CKD and CVD progression.

It has been estimated that approximately 6% of the general population has elevated albuminuria, and that the majority of these subjects are not known yet with this abnormality. Among these subjects, many have hypertension, hyperlipidemia, diabetes and/or impaired kidney function, that often is also not known yet. Early detection of elevated albuminuria may be important because it gives the opportunity to invite subjects that test positive for further screening for CKD and CVD risk factors. Thus these risk factors for CKD and CVD progression could be treated in an early stage.

Population screening for albuminuria could be justified according to the WHO criteria of Wilson and Jungner , because CKD has important consequences for subjects, the course of the disease is initially symptomless, and there are treatment methods available. However, implementation research to validate screening the general population for albuminuria and related health consequences is lacking, as are cost-effectiveness studies.

In the current study the aim is to develop a home-based screening technique for detecting elevated albuminuria. Two screening methods will be investigated, and yield and cost-effectiveness of these screening methods will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 80 years.
* Living in the municipality of Breda, The Netherlands.
* Not institutionalised.

Exclusion Criteria:

* Younger than 45 years or older than 80 years.
* Not living in the municipality of Breda, The Netherlands.
* Institutionalised.

A random sample of 15.032 subjects will be drawn from the population aged 45-80 years from the municipality of Breda by the Dutch Central Bureau for Statistics (CBS).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15032 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Participation rate of the screening (i.e. home-based screening, elaborate screening and overall screening program) | Screening period of 6 months.
  The participation rate is defined as the number of persons completing the albuminuria screening (i.e. returning the first PeeSpot urine device or scanned the first ACR | EU urine test strip with use of the app, and in case of an ACR >30 mg/g in this initial test, also completing the a confirmatory albuminuria screening tests), elaborate screening and overall screening program relative to the invited number of individuals.
The yield of albuminuria screening. | Screening period of 6 months.
  These are twofold. First, the yield of the home-based screening is defined as the number of persons who test positive for albuminuria (at least 2 tests positive) relative to the number of persons participating in the corresponding arm (=per-protocol analysis) and of all invited persons in the corresponding arm (intention-to-screen analysis).
  Second, the yield of the elaborate screening is defined as the number of subjects with increased albuminuria (defined as ACR >30 mg/g) with newly diagnosed and/or poorly controlled CVD and CKD risk factors. These risk factors, which will be assessed during the elaborate screening, include hypertension, diabetes mellitus, hyperlipidemia, impaired kidney function.
Cost-effectiveness of the screening. | 6 months follow-up after screening period.
  Incremental cost-effectiveness ratio (ICER) in euro per QALY gained for the two screening methods;

SECONDARY OUTCOMES:
GP follow-up rate. | Screening period of 6 months.
  Number of persons completing the complete study (ACR testing, elaborate screening when invited, and visiting GP when recommended) relative to the number of referred individuals.
Characteristics of responders. | Screening period of 6 months.
  Information on (differences in) characteristics of the responders of the two screening methods (PeeSpot vs. ACR | EU) including differences in age, sex, educational level, estimated social economic status (based on data of Statistics Netherlands, providing estimated social economic status based on postal codes), medication use, and history of disease
Characteristics of non-responders. | Screening period of 6 months.
  Information on (differences in) characteristics of the non-responders of the two screening methods (PeeSpot vs. ACR | EU) including differences in age, sex, and estimated social economic status.
Usability scores of the two screening methods. | 6 months follow-up after screening period.
  Usability of both tests assessed by questionnaire in the participants with a confirmed positive test and in a subgroup of participants with a negative test.

OTHER OUTCOMES:
Appropriate treatment after elaborate screening. | 6 months follow-up after screening period.
  Evaluate whether the subjects who participated the elaborate screening and in which abnormalities were found (hypertension, diabetes, hypercholesterolemia, impaired renal function) did visit their general practitioner for start of appropriate treatment (lifestyle advice and/or medication).
Information regarding sensitivity and specificity of the home-based screening tests | Screening period of 6 months.
  Information on rate of false-negative and -positive tests for both screening methods (PeeSpot vs. ACR | EU).
Optimal cut-off value of albuminuria. | 6 months follow-up after screening period.
  To investigate which cut-off value of albuminuria should be used in the screening to render the most effective screening.
Optimal age range for albuminuria screening. | 6 months follow-up after screening period.
  Investigate the most effective age range for albuminuria screening.
Role of health literacy in albuminuria screening. | 6 months follow-up after screening period.
  The role of health literacy (assessed by questionnaire) in participating in the screening program and by obtaining appropriate treatment by the GP.

CONTACTS AND LOCATIONS:
Overall Officials: Ron T Gansevoort, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Mil D, Kieneker LM, Evers-Roeten B, Thelen MHM, de Vries H, Hemmelder MH, Dorgelo A, van Etten RW, Heerspink HJL, Gansevoort RT. Participation rate and yield of two home-based screening methods to detect increased albuminuria in the general population in the Netherlands (THOMAS): a prospective, randomised, open-label implementation study. Lancet. 2023 Sep 23;402(10407):1052-1064. doi: 10.1016/S0140-6736(23)00876-0. Epub 2023 Aug 16. PMID 37597522
- [Derived] van Mil D, Kieneker LM, Evers-Roeten B, Thelen MHM, de Vries H, Hemmelder MH, Dorgelo A, van Etten RW, Heerspink HJL, Gansevoort RT. Protocol for a randomized study assessing the feasibility of home-based albuminuria screening among the general population: The THOMAS study. PLoS One. 2022 Dec 22;17(12):e0279321. doi: 10.1371/journal.pone.0279321. eCollection 2022. PMID 36548281